CLINICAL TRIAL: NCT00487669
Title: Phase II Study of the Combination of Paclitaxel Poliglumex (CT-2103, Xyotax) and Pemetrexed (Alimta) for the Treatment of Patients With Advanced Non-small Cell Lung Cancer.
Brief Title: Phase II Study of Combination of Paclitaxel Poliglumex and Alimta for Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-0433
Record Dates: First submitted 2007-06-14; First posted 2007-06-18 (Estimated); Results first posted 2014-01-09 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2013-11

CONDITIONS: Advanced Non-small Cell Lung Cancer
Keywords: paclitaxel poliglumex; xyotax; alimta; advanced non-small cell lung cancer
MeSH Terms: interventions — paclitaxel poliglumex; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel Poliglumex with Pemetrexed (Experimental): The first 6 eligible patients will be enrolled at a dose of 135 mg/m2 paclitaxel poliglumex in combination with 500 mg/m2 of pemetrexed. Patients who experience disease progression without dose-limiting adverse events after the initial cycle will be replaced. Dose escalation to the next dose level can occur provided that no more than 1 of 6 patients experience in initial dose limiting toxicity (IDLT) following 2 cycles of therapy. If ≥ 2 of 6 patients experience IDLTs at the 135 mg/m2 dose, the maximally tolerated dose (MTD) was surpassed and the study will be discontinued.
  Interventions: Drug: paclitaxel poliglumex, pemetrexed

INTERVENTIONS:
Drug: paclitaxel poliglumex, pemetrexed — The first 6 eligible patients will be enrolled at a dose of 135 mg/m2 paclitaxel poliglumex in combination with 500 mg/m2 of pemetrexed. Patients who experience disease progression without dose-limiting adverse events after the initial cycle will be replaced. Dose escalation to the next dose level can occur provided that no more than 1 of 6 patients experience in initial dose limiting toxicity (IDLT) following 2 cycles of therapy. If ≥ 2 of 6 patients experience IDLTs at the 135 mg/m2 dose, the maximally tolerated dose (MTD) was surpassed and the study will be discontinued
  Other Names: Xyotax; Alimta

SUMMARY:
This is a non-randomized, single-arm, single-institution, open label, two-stage phase II and dose-ranging study designed to evaluate the efficacy and safety of paclitaxel poliglumex in combination with pemetrexed in patients with advanced stage IIIB or stage IV NSCLC.

DETAILED DESCRIPTION:
Primary objective

To evaluate the overall response rate (complete plus partial responses by RECIST criteria) to the combination of paclitaxel poliglumex and pemetrexed as therapy in patients with advanced NSCLC.

Secondary Objectives

To evaluate the safety and adverse event profile of the combination of paclitaxel poliglumex and pemetrexed as therapy in patients with advanced NSCLC.

To evaluate the duration of response, time to progression, and overall survival of advanced NSCLC treated with the combination of paclitaxel poliglumex and pemetrexed.

To compare the overall response rate using three-dimensional reconstruction of target lesions by Medical Metrx Solutions (MMS) and RECIST criteria.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of locally advanced and/or metastatic NSCLC (Stage IIIB or IV).
* Bidimensionally measurable lesions or unidimensionally evaluable lesions.
* Age ≥ 18 years.
* At least one measurable target lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST), which has not been previously treated with local therapy (e.g. radiation therapy, chemoembolization, surgery, etc.).
* May have received prior chemotherapy (including taxanes) for advanced NSCLC.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Life expectancy > 12 weeks.
* No active infections.
* Adequate liver and bone marrow function.
* AST<2.5 x ULN, bilirubin <1.5x ULN, alkaline phosphatase<2.5 x ULN (unless bone origin and no liver metastases are documented).
* ANC ≥ 1,500/uL, platelet count ≥ 100,000/uL.
* Normal PT and PTT.
* Bisphosphates initiated prior to study entry will be permitted. However, initiation of bisphosphonates following study entry is not permitted.
* Patients with treated brain metastases must be neurologically stable.
* At least 3 weeks since last chemotherapy and recovered from treatment-related adverse events ≤ grade 1.
* At least 3 weeks since prior radiation and recovered from treatment-related adverse events ≤ grade 1.
* Women of childbearing potential are eligible for the study, provided they have a negative serum or urine pregnancy test within three days of study entry, and an adequate method of contraception is used. Acceptable methods of birth control include barrier methods (condoms, diaphragms with spermicide) or intrauterine devices (IUD). Women whose sole sexual partner is infertile, or who are not sexually active, are also eligible.
* Able to provide written informed consent.

Exclusion Criteria:

* Grade 2 or greater peripheral neuropathy, according to the National Cancer Institute-Common Toxicity Criteria.
* Clinically significant pleural, pericardial or abdominal effusions.
* Untreated brain metastases.
* Patients with previously diagnosed brain metastases will be eligible if they are neurologically stable and have recovered from the effects of radiotherapy or surgery (≤ grade 2).
* Patients with brain metastases must have at least one other site of measurable disease.
* Concurrent radiotherapy.
* Other concurrent cancer treatment-related investigational agent. Investigational supportive care medications are permitted.
* Concurrent treatment with unfractionated heparin or warfarin.
* History of radiotherapy encompassing greater than 50% of the marrow-bearing skeleton.
* Prior bone marrow or stem cell transplant.
* History of other active malignancy within the last year requiring chemotherapy, not including curatively-treated carcinoma in situ of the cervix, or non-melanoma skin cancer (basal cell carcinoma or squamous cell carcinoma).
* Uncontrolled infection.
* Active bleeding, or history of bleeding requiring transfusion within 2 weeks of study entry.
* Active cardiac disease, as defined as:
* Current history of uncontrolled or symptomatic angina.
* History of arrhythmias requiring medications or clinically significant arrhythmias, with the exception of uncomplicated atrial fibrillation.
* Myocardial infarction < 6 months from study entry.
* Any other cardiac conditions, which in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R Rigas, MD, Principal Investigator — Norriss Cotten Cancer Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Paclitaxel Poliglumex With Pemetrexed
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Paclitaxel Poliglumex With Pemetrexed
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Overall Response Rate (Complete Plus Partial Responses by RECIST Criteria) to the Combination of Paclitaxel Poliglumex and Pemetrexed as Therapy in Patients With Advanced NSCLC.
Time Frame: CT or MRI scans of the chest will be obtained after every 2 cycles (6-week intervals +/- 7 days)
Measure: Number; unit: participants
Groups:
- Level 1: The first 6 eligible patients were enrolled at a dose of 135 mg/m2 of paclitaxel poliglumex administered intravenously over 10-20 minutes followed by 500 mg/m2 of pemetrexed administered intravenously over 10 minutes every 3 weeks.
- Level 2: Dose escalation to the next dose level, paclitaxel poliglumex at 175 mg/m2 and pemetrexed at 500 mg/m2, occurred when no more than 1 of 6 patients experience initial dose limiting toxicity (IDLT) following 2 cycles of therapy on the first dose level. If ≥ 2 of 6 patients experience IDLTs, the maximally tolerated dose (MTD) would have been surpassed and the study stopped.
Arm/Group | Level 1 | Level 2
Number analyzed (Participants) | 6 | 6
participants
  Stable Disease | 5 | 4
  Progressive Disease | 1 | 2

2. Secondary Outcome: Time to Progression
Time Frame: time from study entry until the first documented sign of progression
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Level 1 | Level 2
Number analyzed (Participants) | 6 | 6
months | 3.8 [1.5 to 9.2] | 2.8 [0.7 to 10.5]

3. Secondary Outcome: Overall Survival
Time Frame: time from study entry until death
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Level 1 | Level 2
Number analyzed (Participants) | 6 | 6
months | 7.7 [3.7 to 21.4] | 8.5 [2.4 to 22.2]

ADVERSE EVENTS:
Arm/Group | Level 1 | Level 2
Serious Adverse Events (participants affected / at risk) | 0/6 | 5/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Level 1 (N=6) | Level 2 (N=6)
Neutropenia Grade 3 (Blood and lymphatic system disorders) | 0 | 2
Neutropenia Grade 4 (Blood and lymphatic system disorders) | 0 | 1
Fatigue Grade 3 (General disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No